CLINICAL TRIAL: NCT03060538
Title: A Phase Ib, Randomized, Blinded, Placebo-Controlled, Multiple Ascending-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Subcutaneous BFKB8488A in Patients With Type 2 Diabetes Mellitus and Patients With Non-Alcoholic Fatty Liver Disease
Brief Title: A Multiple Ascending Dose Study to Evaluate Safety and Tolerability of BFKB8488A in Participants With Type 2 Diabetes Mellitus and Participants With Non-Alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC39547
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Multiple Ascending Dose BFKB8488A (Experimental): Participants will be randomized to receive BFKB8488A. When adequate safety data are available, a review will be done for all participants to make a dose-escalation or dose and/or regimen modification decision. This will be repeated for each cohort.
  Interventions: Drug: BFKB8488A
- Placebo (Placebo Comparator): Participants will receive BFKB8488A-matching placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BFKB8488A — Administered subcutaneously starting on Day 1 and according to dosing schedule.
  Other Names: RO7040551
  Arms: Multiple Ascending Dose BFKB8488A
Other: Placebo — Administered subcutaneously starting on Day 1 and according to dosing schedule.
  Arms: Placebo

SUMMARY:
This is a Phase Ib, randomized, blinded, placebo-controlled, multiple ascending-dose study of the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) effects of BFKB8488A in participants with Type 2 diabetes mellitus (T2DM) and participants with non-alcoholic fatty liver disease(NAFLD). A maximum of approximately 160 participants will be enrolled across multiple sites in the United States. Participants will be randomly assigned to receive study drug (active BFKB8488A or placebo). The study will consist of a screening period (up to 8 weeks), a 12-week treatment period, and a 6-week follow-up period. Participants may come to clinic for an optional pre-screening visit.

ELIGIBILITY:
Inclusion Criteria:

For T2DM Cohort only:

* Body mass index (BMI) ≥ 27 kg/m2 and ≤ 40 kg/m2.
* A confirmed diagnosis of Type 2 diabetes ≥ 6 months at screening
* Current stable treatment (at least 3 months) for diabetes
* Hemoglobin A1c (HbA1c) ≥ 6.8% and ≤ 9.0%.
* For women of childbearing potential, agreement to remain abstinent or use reliable contraception during treatment period and for at least 42 days after last dose of study drug
* For men, agreement to remain abstinent or use reliable contraception and agree to refrain from donating sperm
* For NAFLD cohort only:
* BMI ≥ 25 kg/m2 and ≤ 40 kg/m2
* At screening, confirmed liver fat by ultrasound OR calculated Liver Fat ≥ 10% using variables from the NAFLD liver fat score
* Hepatic steatosis on magnetic resonance imaging (MRI; ≥ 10% average liver proton density fat fraction [PDFF]) prior to randomization.

Exclusion Criteria:

* Pregnant, lactating, or intending to become pregnant within 42 days after the last dose of study drug is administered
* Suspected or confirmed diagnosis of Type 1 diabetes
* Significant cardiac disease
* Any psychiatric illness that increases the risk of participation in the study
* History of severe allergic, anaphylactic, or other hypersensitivity reactions, or severe systemic bacterial, fungal, or parasitic infections
* Poor peripheral venous access
* Received blood products within 2 months before dosing
* Donation or loss of blood within 30-56 days prior to study drug administration
* Positive for hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody
* Liver enzymes greater than acceptable limits
* History of eating disorders or surgical procedures for weight loss
* Active participation in a structured weight loss or dietary program
* Treatment with investigational therapy or exposure to any biological therapy
* Illicit drug use, marijuana use, or alcohol abuse
* Current use of more than one pack of cigarettes a day or equivalent nicotine- containing products
* Any serious medical condition or abnormality in clinical laboratory tests

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2017-03-05 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AE) | Up to 18 weeks following first dose administration
  An adverse event is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution.

SECONDARY OUTCOMES:
Serum BFKB8488A Concentration | On multiple days during treatment period and follow-up (up to 18 weeks following first dose administration)
Change from Baseline in Percentage of Participants with Anti-Therapeutic Antibodies (ATAs) | On multiple days during treatment period and follow-up (up 18 weeks following first dose administration)
  Participants are considered to be ATA positive if they are ATA negative at baseline but develop an ATA response following study drug administration (treatment-induced ATA response), or if they are ATA positive at baseline and at least one post-baseline samples if above acceptable limits. The number and percentage of ATA-positive and ATA-negative participants will be summarized by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- United States (17):
  - Pinnacle Research Group Cullman, Anniston, Alabama
  - Pinnacle Research Group; Llc, Central, Anniston, Alabama
  - Southern California Research Center, Inc., Coronado, California
  - Stanford Health Care, Stanford, California
  - Diabetes Research Center, Tustin, California
  - MD Clinical, Hallandale, Florida
  - Premier Research Associate, Inc, Miami, Florida
  - Agile Clinical Research Trials, Atlanta, Georgia
  - MidWest Clinical Research, Overland Park, Kansas
  - Hassman Research Institute, Berlin, New Jersey
  - Carolina Research Center at Jones Family Practice, Shelby, North Carolina
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - Clinical Trials of Texas Incorporated, San Antonio, Texas
  - Northeast Clinical Research of San Antonio LLC, San Antonio, Texas
  - Consano Clinical Research, Shavano Park, Texas
- inVentiv Health Clinical, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Wong C, Dash A, Fredrickson J, Lewin-Koh N, Chen S, Yoshida K, Liu Y, Gutierrez J, Kunder R. Fibroblast growth factor receptor 1/Klothobeta agonist BFKB8488A improves lipids and liver health markers in patients with diabetes or NAFLD: A phase 1b randomized trial. Hepatology. 2023 Sep 1;78(3):847-862. doi: 10.1002/hep.32742. Epub 2022 Sep 12. PMID 35993161